CLINICAL TRIAL: NCT04270214
Title: Conversion and Optimization of Dysport for Cervical Dystonia
Brief Title: Conversion to Dysport in CD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Mandar Jog, Movement disorders neurologist, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115308
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Cervical Dystonia
Keywords: botulinum toxin type A
MeSH Terms: conditions — Torticollis | interventions — abobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dysport (Other): Single arm study, all participants will receive Dysport injections
  Interventions: Drug: Dysport Injectable Product

INTERVENTIONS:
Drug: Dysport Injectable Product — Dysport injections optimized using kinematics
  Other Names: abobotulinumtoxinA

SUMMARY:
The first line of therapy for cervical dystonia patients is botulinum toxin injections, however injection parameter determination and optimization are challenging for physicians to do. In addition, some patients receiving this treatment long-term experience short duration of relief. Thus, Dysport (Ipsen Biopharmaceuticals), another BoNT-A formulation, may increase the duration of clinical benefit. The objective of this study is to compare the wearing off time of their original BoNT-A formulation (same injection parameters for at least 3 cycles) and the optimized treatment of Dysport (after 2 injection cycles). Ideally, the clinical benefits should last 2.5 - 3 months as injections are administered every 3 months. Conversion to Dysport will be conducted and optimization of Dysport dosing will be done using our sensor-technology assessment. It is unclear whether there are differences in the neurophysiological effects between BoNT-A formulations, such as blocking spinal afferent signals from proprioceptive mechanoreceptors of the injected muscles contributing to CD or the modulation of cortical activity [8]. The underlying pathophysiology of impaired motor control in CD is theorized to be caused by abnormal somatosensory processing that affects proprioceptive and tactile function [8]. By altering the processing of proprioceptive signals from the muscles to the cortical somatosensory-motor areas, proprioceptive perception can be modulated and possibly normalize activity of the somatosensory-motor areas in CD. Thus, it is hypothesized that BoNT-A may indirectly modulate these cortical pathways and Dysport may have a longer modulatory effect to produce a longer lasting clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cervical dystonia
* Patients experiencing early waning off (benefit for up to 8 weeks) of their current BoNT-A treatment (stable for at least 3 treatments)
* Only those that want to switch to Dysport will be included.
* No prior exposure to Dysport
* Able to come for multiple visits
* Patient's injection parameters are stable for ≥3 cycles
* Patient can provide written consent

Exclusion Criteria:

* Unable to come for study visits

  1. Receiving BoNT-A for other indications (e.g. upper limb tremor)
  2. if you have a history of seizures.
  3. Pregnancy or Nursing: If you are pregnant then you ARE NOT ELIGIBLE FOR THIS STUDY. Please notify the research team if you are presently pregnant or if you are attempting to become pregnant or if you become pregnant at any time during the course of the study. A researcher will ask you about pregnancy at every study visit. If you are nursing, you ARE NOT ELIGIBLE FOR THIS STUDY. Please notify the researcher. Results from a pregnancy test will confirm your pregnancy status.
  4. Other Muscle/Nerve diseases: If you have a disease called Myasthenia Gravis or Amyotrophic Lateral Sclerosis (ALS or Lou Gehrig's disease) then you ARE NOT ELIGIBLE FOR THIS STUDY. Please notify the research team if you have these conditions.
  5. Previous side effects to botulinum toxin: If you have had a previous allergic reaction or side effect to botulinum toxin then you MAY NOT BE ELIGIBLE FOR THIS STUDY. Pease notify the research team if you have had a previous reaction/side effects from injection of botulinum toxin.
  6. Myotomy or denervation surgery: If you have had previous surgery for a myotomy or denervation of the neck or shoulder region then you ARE NOT ELIGIBLE FOR THIS STUDY. Please notify the research team if you have ever had these surgeries.
  7. allergy to cow's milk protein

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
waning effect | within 12 weeks of treatment
  telephone call report of when participant perceives benefit of treatment is wearing off

SECONDARY OUTCOMES:
objective measures of CD severity | 4-weeks and 12-weeks post-treatment
  Kinematic sensor technology is used to measure CD symptoms (neck pulling and/or tremor). Sensors coupled with computer-assisted analysis can measure degrees of deviation from neutral head/neck position and angular root mean square tremor/dystonic jerks amplitude in each plane of motion (vertical, lateral, rotational).
changes in TMS measures | 4-weeks and 12-weeks post-treatment
  changes in brain activity (inhibitory and excitatory pathways) using paired pulse TMS. Using established techniques
visual-motor performance | 4-weeks and 12-weeks post-treatment
  speed, reaction time and accuracy in completing upper limb target reaching choice tasks using a robotic haptic device

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No